CLINICAL TRIAL: NCT03036215
Title: Tailored Self-Management of TMD Pain Using Health Information Technology
Brief Title: Tailored Self-Management of Temporomandibular Disorders (TMD) Using Health Information Technology
Acronym: TMDPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5U01DE025609-02 (NIH)
Record Dates: First submitted 2017-01-18; First posted 2017-01-30 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2017-01

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome

STUDY DESIGN:
Intervention Model Description: The pilot study design is a 2-arm randomized clinical trial to test the methods that will be used in a future proposal for a full-scale multi-site clinical trial. The two aims include: 1) evaluate the feasibility of methods to conduct a full-scale multi-site randomized clinical trial comparing the PACT self-management with usual self-care for TMD and, 2) estimate the parameters needed to plan for a larger multi-site trial including the effect size and standard deviation for primary outcomes of pain and function. A traditional self-care control arm is added to determine the acceptability of randomization and the feasibility of collecting baseline and follow-up data from a traditional care control arm for the full-scale study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Self-Care Control Arm (No Intervention): Traditional self-care includes focusing on rest and healing through changes in chewing, diet, heat/cold, over the counter analgesics, and reducing strain from oral and sleeping habits. Participants will also participate in usual care from the dentist such as a splint or anti-inflammatory medications. Participants will complete follow-up measures at 8-weeks (post-intervention) and at 16-weeks (2 months after program end). .
- PACT Experimental Arm (Experimental): If selected for the PACT care arm, participant will be prompted to complete a self-management program, entitled Personalized Activated Care and Training (PACT) that is a tailored 8-week progressive web-based training program supported by a health coach to enhance understanding, compliance, and success in improving TMD pain. Participant will also participate in usual care from the dentist such as a splint or anti- inflammatory medications.Participant will complete follow-up measures at 8-weeks (post-intervention) and at 16-weeks (2 months after program end).
  Interventions: Behavioral: PACT Experimental Arm

INTERVENTIONS:
Behavioral: PACT Experimental Arm — The study will employ a self-management program, entitled Personalized Activated Care and Training (PACT) that is a tailored 8-week progressive web-based training program supported by a health coach to enhance understanding, compliance, and success in improving TMD pain. The program provides 8 weeks of structured didactic and experiential training on exercises and cognitive- behavioral training to reduce risk factors that contribute to delayed recovery and enhance protective factors that have evidence of improving TMD pain.
  Arms: PACT Experimental Arm

SUMMARY:
The purpose of this pilot project is to determine the feasibility and acceptability of proposed methods for a subsequent clinical trial of a tailored self-management program (PACT) designed to decrease pain in participants with temporomandibular disorders (TMD). The PACT program is a personalized program of exercise and behavioral changes implemented through a web-based program supported by a health coach. For this feasibility and acceptability study, 80 adults with TMD pain will be randomized either to the PACT program or to traditional self-care.

DETAILED DESCRIPTION:
The primary study objectives of the PACT study are two-fold:

1. Evaluate the feasibility of methods to conduct a full-scale multi-site randomized clinical trial comparing PACT self-management with traditional self-care for TMD. The study will also evaluate strategies to: identify, recruit, consent, and enroll eligible subjects into both groups meeting target goal; evaluate adherence to intervention and identification of barriers; evaluate adherence to outcomes assessment, and evaluate the on-line web-site functionality and acceptability.
2. To demonstrate ability to accurately capture outcome measures to be used in the multi-site study.

Primary study objective: Recruitment is measured through achievement of target sample, number of patients identified that meet eligibility criteria, and number (%) of subjects consenting compared with total contacted.

Intervention adherence is measured by: number of participants enrolled in both groups, number of participants accessing on-line materials, completion of practice logs, and identification of self-reported barriers of participation in self-care. Outcome adherence is measured by the number of participants who complete the baseline assessment, complete the two and four month follow-up assessments, complete the program evaluation, and complete qualitative post-study interview. Website acceptability is measure by identification of problems and barriers during use and quality and ease of use at the post-intervention evaluation.

Second objective: Efficacy of the program is measured by self-reported outcome assessments. The primary outcomes include TMD symptoms, jaw functioning, and emotional functioning. Secondary outcomes measures include symptom severity with the temporal aspects of pain, pain interference, and patient ratings of improvement. Additional information on mediators and modifiers will also be gathered to help inform the how and why the intervention has an effect. Mediators will be measured to identify factors that help explain why PACT may have an effect including self-efficacy, patient activation, exercise level, sleep quality, and social support. Contextual process factors to identify in whom the intervention does and does not work include disability status, catastrophizing, depression, repetitive strain from oral habits, and perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, an individual must meet all of the following criteria:

  * Age 18 or older
  * Able and willing to access the internet on a regular basis
  * Able to read and speak English
  * Be willing to comply with all study procedures:

    1. Randomly assigned to either arm of the study
    2. Be available for the duration of the study
    3. Complete study data collection forms
    4. Reachable by phone and able to participate in weekly phone coaching calls if randomized to the PACT arm
  * Have a diagnosis of TMD pain using a self-report screener. These questions include;

    1. In the last 30 days, which of the following best describes any pain in your jaw or temple area on either side?
    2. In the last 30 days, have you had pain or stiffness in your jaw on awakening?
    3. In the last 30 days, did the following activities change any pain (that is, make it better or make it worse) in your jaw or temple area on either side? Chewing hard or tough food, Opening your mouth or moving your jaw forward or to the side, Jaw habits such as holding teeth together, clenching/grinding, or chewing gum, or other jaw activities such as talking, kissing, or yawning
  * Frequency of TMD pain more than once a week with pain in the past 6 months
  * Electronically sign an informed consent form

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  * Currently participating in any other TMD and temporomandibular joint (TMJ) related studies
  * Major disk disorder that requires opioids or surgery for TMD pain
  * Serious medical condition that might interfere with or prohibit participation in an online program or pregnancy
  * Treatment for a mental health disorder or substance abuse in the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. Fricton, DDS, Principal Investigator — HealthPartners Institute; Robin R. Whitebird, PhD, MSW, Principal Investigator — University of St Thomas , School of Social Work
Locations (1):
- HealthPartners Clinic, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional Self-Care Control Arm: Traditional self-care focuses on rest and healing through changes in chewing, diet, heat/cold, over the counter analgesics, and reducing strain from oral and sleeping habits. Participants in the traditional arm may also be receiving usual care from their dentist such as a splint or anti-inflammatory medications. They will complete follow-up measures at 8-weeks (post-intervention) and at 16-weeks (2 months after program end).
- PACT Experimental Arm: Participants enrolled in the experimental arm are prompted to complete a self-management program, Personalized Activated Care and Training (PACT), The program provides 8 weeks of structured didactic and experiential training on exercises and cognitive- behavioral training to reduce risk factors that contribute to delayed recovery and enhance protective factors designed to improve TMD pain. Participants also complete follow-up measures at 8-weeks (post-intervention) and at 16-weeks (2 months after program end). These participants are also supported by a health coach.
Period: Overall Study
Arm/Group | Traditional Self-Care Control Arm | PACT Experimental Arm
Started | 41 | 39
Completed | 39 | 36
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- PACT Experimental Arm: PACT Experimental Arm: The study employs a self-management program, entitled Personalized Activated Care and Training (PACT) that is a tailored 8-week progressive web-based training program supported by a health coach to enhance understanding, compliance, and success in improving TMD pain. The program provides 8 weeks of structured didactic and experiential training on exercises and cognitive- behavioral training to reduce risk factors that contribute to delayed recovery and enhance protective factors that have evidence of improving TMD pain.
- Total: Total of all reporting groups
Arm/Group | Traditional Self-Care Control Arm | PACT Experimental Arm | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (15.1) | 46 (17.1) | 47.5 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 38 | 38 | 76
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 36 | 34 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 41 | 39 | 80
Graded Chronic Pain Severity [Mean (Standard Deviation); unit: units on a scale] — Pain Intensity is a O-100 score derived from questions 1-3:
  Mean (Pain Right Now, Worst Pain, Average Pain) x 10; Item Scale is from 0=No pain to 10=Pain as bad as it could be
  units on a scale | 50 (15) | 50 (17.6) | 50 (16)
Graded Chronic Pain interference [Mean (Standard Deviation); unit: units on a scale] — Graded Chronic Pain Interference subscale:
  Interference Score is a O-100 score derived from 3 questions:
  Mean (Daily Activities, Social Activities, Work Activities) x 10; Scale 0=no interference up to 10=unable to carry on activities
  units on a scale | 26.6 (23.7) | 23 (21.3) | 24.9 (22.5)
Jaw Functioning [Mean (Standard Deviation); unit: units on a scale] — Level of limitation during the last 30 days. Scale 0-10 of drink, Soft food, Swallow, Talk, Smile, Chew, Yawn, Hard food. JAW FUNCTIONING 8 items R:0-80; Item scale: 0 = No limitation up to 10=Severe limitation
  units on a scale | 24.5 (18.9) | 19.4 (14) | 22 (16.8)

OUTCOME MEASURES:

1. Primary Outcome: Assessing Graded Chronic Pain Severity Evaluation Feasibility of the PACT Program
Description: Measure: Graded Chronic Pain Scale (GCPS) with mean intensity ratings for reported current, worst, and average pain. 3 items: Scale 0-100 (100 most severe)
Time Frame: Change from baseline to 16 weeks post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Traditional Self-Care Control Arm | PACT Experimental Arm
Number analyzed (Participants) | 39 | 36
units on a scale | -12 (16.8) | -19 (16)
Statistical Analysis 1: Comparison: Traditional Self-Care Control Arm vs PACT Experimental Arm; Pilot study, no power analysis applicable; no statistical test; Test type: Other; Mean Difference (Net) = -7

2. Primary Outcome: Assessing Change in Jaw Functioning
Description: Jaw Functional Limitation Scale (JFLS-8) identifies daily activities interfered with by jaw pain - 8 items Scale 0-80 (80 more severe)
Time Frame: Change from baseline to 16 weeks post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Traditional Self-Care Control Arm | PACT Experimental Arm
Number analyzed (Participants) | 39 | 36
units on a scale | -7.9 (14.9) | -6.9 (19.6)
Statistical Analysis 1: Comparison: Traditional Self-Care Control Arm vs PACT Experimental Arm; Pilot study; no statistical test run; Test type: Other — pilot study; no statistical test performed; Mean Difference (Net) = 1

3. Secondary Outcome: Graded Chronic Pain Interference
Description: Assessment of graded Chronic Pain Interference - Scale (0-100); 0 = lowest pain interference 100 = highest pain interference. If findings in negative values = improvement; positive values = worsening condition.
Time Frame: Change from baseline to 16 weeks post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Traditional Self-Care Control Arm | PACT Experimental Arm
Number analyzed (Participants) | 39 | 36
units on a scale | -5.8 (20.7) | -11 (17.2)
Statistical Analysis 1: Comparison: Traditional Self-Care Control Arm vs PACT Experimental Arm; Pilot study; no statistical test for significance run; Test type: Other; Mean Difference (Net) = -5.2

ADVERSE EVENTS:
Time Frame: through study completion; an average of 16 weeks.
Groups:
- PACT Experimental Arm: PACT intervention employs a self-management program, entitled Personalized Activated Care and Training (PACT) that is a tailored 8-week progressive web-based training program supported by a health coach to enhance understanding, compliance, and success in improving TMD pain. The program provides 8 weeks of structured didactic and experiential training on exercises and cognitive- behavioral training to reduce risk factors that contribute to delayed recovery and enhance protective factors that have evidence of improving TMD pain.
Arm/Group | Traditional Self-Care Control Arm | PACT Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03036215/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03036215/SAP_001.pdf
  • Informed Consent Form (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT03036215/ICF_002.pdf